CLINICAL TRIAL: NCT00438074
Title: A Pilot Study To Evaluate the Effectiveness of Pulsed Time-Domain Optical Spectroscopy for Monitoring the Responses in Neoadjuvant Treatments of Locally-Advanced Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: ART Advanced Research Technologies Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Gregory Czarnota, Dr., Sunnybrook Health Sciences Centre
Other Study IDs: 186-2006
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Diffuse Optical Spectroscopy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This study will investigate optical tissue characteristics as a function of neoadjuvant breast cancer treatment. Our objective in this pilot study will be to identify diffuse optical spectroscopy parameters that change with treatment and that may correlate with pathological response. The ultimate goal is to use such parameters ultrasound as an early predictor of pathological partial or complete response in women with locally advanced breast cancer receiving treatment with neoadjuvant treatments such as chemotherapy or neoadjuvant combined modality chemotherapy and radiotherapy.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy for females in North America. Around 5-15% of the estimated 200,000 new cases diagnosed each year will present with locally advanced breast cancer (LABC) (The definition of what constitutes "LABC" is complex and variable. Clinically these tumours are usually considered to be those greater than 5cm in size and/or extend beyond the breast tissue into the surrounding skin or muscle. Patients with matted axillary lymph nodes (N2) or internal mammary nodes (N3) or ipsilateral supraclavicular lymph node involvement are also considered to have LABC. In view of the extensive nature of these tumours at presentation, women with LABC have a poor outcome in terms of both local and systemic recurrence. Standard treatment for these patients is usually neoadjuvant systemic (chemotherapy or less frequently endocrine therapy) followed by surgery and radiotherapy. Patients who have hormone receptor positive tumours will then receive endocrine therapy. With the use of multidisciplinary therapy, 10-year disease free survival rates of 50% for Stage IIIA and 33% for Stage IIIB disease have been reported.

The impetus for undertaking this study is that we are searching for imaging methods that could potentially serve as surrogate indicators of pathological response. One such modality that we wish to investigate as it may be ultimately useful in this patient population is diffuse optical spectrometry. This modality depends on differentiating oxygenated from deoxygenated tissue but is also sensitive to other changes in tissue characteristics. It has been used before in proof-of-principle studies differentiating benign from malignant disease but we hypothesize that it may be more useful in terms of monitoring tumour responses to treatment. This is a non-invasive imaging modality that is easy to administer and relatively inexpensive.

ELIGIBILITY:
Inclusion Criteria:

* Locally Advance Breast Cancer
* Subjects must give appropriate written informed consent prior to participation in the study;
* Subjects must be able and willing to comply with the safety procedures during the Scanning Period;
* Subjects must be women of between 20 and 80 years of age, inclusive, on the day the Informed Consent Form is signed;
* Subjects must be women who will be receiving neoadjuvant radiation therapy and/or chemotherapy for locally-advanced breast cancer.
* Subjects of childbearing potential must be using an acceptable method of birth control. Subjects not of childbearing potential are defined as either surgically sterile or post-menopausal. Post-menopausal women are defined as those women with a documented menstruation cessation for 12 consecutive months prior to signing the Informed Consent Form

Exclusion Criteria:

* Subjects with a past medical history of abnormalities, significant injury, or medical or surgical procedures (e.g.,silicone/saline implants) involving either breast, exclusive of the lesion at issue;
* Subjects with any dermatologic abnormalities (including tattoos, open sores, or breached skin) involving either breast;
* Subjects with a current or past medical history of connective tissue disease;
* Subjects who are pregnant or lactating;
* Subjects with an implanted electronic device such as a cardiac pacemaker, defibrillator, or neurological stimulator;
* Subjects with a history or expectation of significant anxiety associated with undergoing diagnostic evaluations;
* Subjects with a history of musculoskeletal disease which may predispose them to discomfort during the Scanning Period;
* Subjects with a known sensitivity to purified water, soybean oil, sucrose, polysorbate 80, oleic acid, EDTA, benzalkonium chloride, FD&C caramel color, butylated hydroxyanisole, and/or sodium hydroxide;
* Subjects with a known sensitivity to low-power infrared radiation (e.g., as a result of a dermatologic condition); and
* Subjects, who, in the opinion of the investigator or clinical research coordinator, may not otherwise be appropriate for inclusion into the study.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who are receiving neoadjuvant chemotherapy or neoadjuvant chemo-radiotherapy for locally-advanced breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2007-02; Primary Completion 2024-05-17 (Estimated); Study Completion 2024-05-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J. Czarnota, Ph.D. M.D., Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada